CLINICAL TRIAL: NCT00877708
Title: Clinical and Microbiologic Characteristics of Cephalosporin-Resistant E. Coli-PITT Protocol
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Yohei Doi, MD, University of Pittsburgh
Other Study IDs: IRB#PRO08100393
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: E Coli Infections
Keywords: E. Coli; isolates
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biologic samples (isolates) will be under the control of the principal investigator of this research project. All samples provided to the investigator are de-identified by the honest broker and will be coded with numbers. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location that only the honest broker has access to. The investigator on this study will keep the samples indefinitely. Samples will be kept in the investigator's laboratory located in Scaife Hall, room 839, 3550 Terrace Street. At no time with the research investigators have access to any patient identifers. Medical record information and bacteria samples from facilities outside of UPMC will be provided to the PI de-identified. At not time will anyone on the research team have access to patient identifiers. All information and bacteria are collected as part of the patient's clinical treatment.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to review patients with E. coli infections at UPMC from September 1, 2008 to August 31, 2010 to determine if these infections have arisen in the community rather than in hospitals or nursing homes and determine their clinical outcomes.

The specific aims of this study are to:

1. Review whether cephalosporin-resistant E. coli infections are hospital-acquired, healthcare-associated or community-associated.
2. Determine the clinical outcome of the patients according to the antibiotics given.

DETAILED DESCRIPTION:
De-identified data will be obtained by the honest broker for the requested time period. In addtion, the honest broker will work with the microbiology laboratory to collect the isolates associated with the de-identified data. All data and samples will be de-identified. De-identified data will be given to the nurse coordinator to complete the case report forms and enter the data into the password protected database and the de-identified isolates will be stored and analyzed on the 8th floor Scaife in Dr. Yohie Doi's laboratory.

ELIGIBILITY:
Inclusion Criteria:

* patients with E. coli infections at UPMC

Exclusion Criteria:

* not meeting entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with E. coli infections at UPMC
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States